CLINICAL TRIAL: NCT06503393
Title: SENOVIE France - Therapeutic Mobility and Breast Cancer
Acronym: SENOVIE
Status: Recruiting | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: The French Institute for Demographic Studies (INED) (Unknown); Saint-Louis Hospital, Paris, France (Other); Centre Hospitalier de Saint-Denis (Other); Centre Hospitalier Intercommunal Robert Ballanger (Other); The French National Cancer Institute (Unknown); The French Collaborative Institute on Migrations (Unknown); Ceped UMR 196 (Unknown); Université Paris Cité (Other)
Responsible Party: Principal Investigator, Clémence Schantz, PhD, Institut de Recherche pour le Developpement
Other Study IDs: IRD_2024_CEPED_SENOVIE
Record Dates: First submitted 2024-06-06; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Female
Keywords: Life-event survey; Observational survey; Breast cancer; Immigrant; Women; Sub-saharan Africa; France; Trajectories; therapeutic itinerary; social inequalities; health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women born in sub-Saharan Africa: Women born in sub-Saharan Africa and diagnosed with breast cancer
- Women born in France: Women born in France and diagnosed with breast cancer

SUMMARY:
Background

In France, there were 61,214 new cases of breast cancer in France in 2023 with an estimated prevalence in 2017 of 913,089 people. It is thus the most common cancer in women, with an incidence that has been increasing since 1990, due both to changes in screening but more recently to a moderate increase in relation to changes in risk factors.

Social inequalities in breast cancer are documented, but there are no data on immigrant women, and there is reason to believe that their trajectories may be different from those of women born in France (characteristics and age of cancer onset, problems of access to care, isolation, etc.).

The SENOVIE France project aims to better understand the impact of breast cancer on the life trajectories of women born in France and women born in sub-Saharan Africa.

Objectives

The SENOVIE France survey aims :

* To understand how breast cancer (diagnosis, treatment, and breast reconstruction) impacts women's lives that are already affected by migration in many spheres (i.e., social consequences of breast cancer on spheres like family or occupation/financial situation).
* To study the therapeutic itineraries (including self-reconstruction) of immigrant women living with breast cancer in the greater Paris area and understand their social determinants.
* To observe how gender can shape women's medical and social outcomes in a migration context.

Methodology

The SENOVIE France survey is a mixed-methods survey with a quantitative and a qualitative component. The quantitative component consists of a quantitative, retrospective, life-event survey carried out among 1000 women living with breast cancer and followed in three health services in the greater Paris area. Women born in France and sub-Saharan Africa will be surveyed. This survey consists of a CAPI patient questionnaire and a biographical grid paper (for the life-event data collection) administered face-to-face by specially trained interviewers, as well as a medical questionnaire completed by the team of the health services concerned. Statistical analyses adapted to longitudinal data will be used to study women's trajectories.

The qualitative component consists of a survey by semi-structured interviews with women living with breast cancer and followed in the greater Paris area. These interviews are the subject of an audio recording and then a pseudonymized transcription. Thematic analyses will be carried out with a comprehensive approach that aims to analyze women's experiences.

Perspectives and expected results

This survey will provide scientific knowledge on the diagnosis, treatment and experience of breast cancer and its impact on the life trajectories of women born in France and sub-Saharan Africa. These results could thus contribute to the improvement of medical and psychosocial care for women living with breast cancer.

DETAILED DESCRIPTION:
Background

In 2023, with 61,214 new cases diagnosed in France, breast cancer accounts for 33% of women's cancers and is the most common cancer in women. With an estimated prevalence in 2017 of 913089 people, studies also suggest an increase in the standardized incidence rate for several years, from 72.8 per 100,000 in 1990 to 99.2 per 100,000 in 2023. This increase is partly explained by the implementation of screening campaigns that promote the early detection of new cases, but also by the presence of risk factors that are responsible for a large proportion of breast cancers.

Studies on social inequalities in the face of breast cancer highlight several realities. Indeed, while breast cancer is considered one of the cancers with a better prognostic life due to the net survival rate of 88% observed five years after diagnosis, studies show that these rates vary by age and that women from lower social classes have a higher risk of death than women from privileged social classes. In addition, although immigrant women, especially those from sub-Saharan Africa, face several health problems and often live in precarious situations in France, few studies have documented the situation of these women with breast cancer compared to women born in France. The few studies carried out highlight inequalities in access to breast cancer screening and a life after breast cancer marked by significant social and administrative precariousness. Thus, it is possible to think that, in the face of breast cancer, the trajectories of women born in sub-Saharan Africa could be different from those of women born in France. For example, it is possible that immigrant women have a different age of cancer onset than non-immigrant women or that they encounter greater difficulties in accessing care.

The SENOVIE France project was designed to fill this knowledge gap. It aims to better understand the impact of breast cancer on the life trajectories of women born in France and women born in sub-Saharan Africa.

Objectives

The SENOVIE France survey aims:

* To understand how breast cancer (diagnosis, treatment, and breast reconstruction) impacts women's lives that are already affected by migration in many spheres (i.e., social consequences of breast cancer on spheres like family or occupation/financial situation).
* To study the therapeutic itineraries (including self- reconstruction) of immigrant women living with breast cancer in the greater Paris area and understand their social determinants.
* To observe how gender can shape women's medical and social outcomes in a migration context.

Methodology

The SENOVIE France survey is a mixed-methods survey with two components: a quantitative component and a qualitative component.

Quantitative component The quantitative component is based on a life event survey, a methodology successfully used in the field of HIV/Hepatitis B among immigrants in the greater Paris area by several members of this research. This innovative methodology has the great advantage of collecting longitudinal data while avoiding attrition which is very frequent in prospective cohorts among disadvantaged populations: women are surveyed one time and are asked retrospectively about their past trajectories. A close-ended question CAPI questionnaire and a biographical grid paper where the interviewer reports key elements and dates will be used for data collection. The biographical grid paper was shown to help to minimise memory biases because the interviewees can use both dates and age to remember the order of events and can place elements in perspective with one another (for example, a woman can ignore at what date she had access to medical insurance, but she would remember it occurred during her second pregnancy). This methodology has shown robustness in tracing back life and health trajectories.

This survey aims to recruit about 1000 women, including 500 women born in France and 500 women born in sub-Saharan Africa. During the twelve months of the data collection, a CAPI patient questionnaire, a biographical grid paper (completed by interviewers recruited and trained by INED) and a medical questionnaire (completed by clinical researchers from partner hospitals) will be used to collect the following data:

The patient questionnaire and the biographical grid include the following modules:

1. retrospective on the whole life (residential history, professional history),
2. history of relationships and children,
3. nationality, arrival in France and stay (for immigrant women),
4. health coverage,
5. violences,
6. breast cancer (diagnosis, treatment, and impact on women's life),
7. Covid period,
8. economic consequences,
9. health, sexuality and well-being.

The collection will be carried out in the context of a face-to-face interview. Within each health services, eligible patients will be identified by the healthcare professional during (or before) the consultation. The survey will be offered by the healthcare professional to all eligible patients. Patients who will agree to participate will be referred to the interviewers. Patients will be able to agree to participate in the survey immediately after their consultation or agree to participate by appointment. Those who will agree to participate by appointment will agree on a date for taking the questionnaire with the interviewers. In both cases, the questionnaire will be administered in the premises of the project's hospital partners (Saint-Louis University Hospital AP-HP ; Delafontaine Hospital Saint-Denis ; Robert Ballanger Hospital Aulnay-sous-Bois) in offices that guarantee the confidentiality of the interview. The individual questionnaires will be entered in real time on an INED secure LimeSurvey server. The biographical grids will be collected on paper before being entered by a dedicated operator on the same LimeSurvey server.

The medical questionnaire contains questions about the characteristics of the cancer and the treatments followed by women. It will be supplemented by hospital staff from partner centres. The entry will be done on the IRD's REDCap secure server.

In terms of statistical analysis, descriptive statistics will be used to precisely describe the medical status, social characteristics, and living conditions of women born in France and women born in Sub-Saharan Africa living with breast cancer in the greater Paris area. These statistics may also be age-standardized if, as expected, women from sub-Saharan Africa are younger than their native-French counterparts.

To measure the social consequences of breast cancer diagnosis and treatments, specific statistical methods for longitudinal data (sequence analysis, Cox models, discreet-time logistic regressions) that allow to take different temporalities into account (time since migration, since diagnosis, since treatment, etc.) will be used. A specific attention will be paid to how healthcare trajectories may have been impacted between 2020 and 2021 by the sanitary crisis, and also to examine whether all women were affected in the same way (missing medical follow-ups, delayed surgeries). Special attention will also be paid to the social determinants and social impacts of breast reconstruction.

Qualitative component

The objective of this qualitative component is to describe in depth the way in which women's health, social and migratory trajectories are articulated, and their involvement in the care of women born in Sub-Saharan Africa in French health services. This section aims to answer the following questions: which immigrant women circulate and under what conditions? What are the challenges and obstacles participants face? What are the administrative, material and social difficulties participants face? What levers can be activated ? To remove these obstacles, which actors can immigrant women rely on? What are the professional, family, conjugal, emotional and physical experiences of these women? To answer these questions, qualitative interviews will be conducted with women born in sub-Saharan Africa. The goal is to carry out about forty interviews in the greater Paris area. The exact number may vary depending on the principle of data saturation. The interviews will be recorded, pseudonymized and transcribed. They will be stored on a secure NextCloud server at Ceped. The interviews will be analyzed with a comprehensive approach that aims to analyze the experiences as they were lived by the participants.

Perspectives and expected results

This research will document the social and health trajectories of women with breast cancer and followed in certain hospitals in the greater Paris area with a comparative aim. It will provide scientific knowledge on the circumstances of cancer diagnosis in women born in France and those born in sub-Saharan Africa, on the experience of the disease and its consequences on different aspects of women's lives (economic, entourage, sexuality, couples, etc.).

This research will raise the awareness of patients' associations and perhaps help them to develop specific lines of action for immigrant women and to lobby political decision-makers to promote their access to care. These results could thus contribute to the improvement of medical and psychosocial care for women living with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or more
* Women who consult in one of the partner hospitals of the study
* For groups 1: women born in a country of sub-Saharan Africa
* For group 2: women born in France
* Have been diagnosed with breast cancer between the 1st of January 2014 and the 31st of December 2020. As data collection will start in 2024, this is to be able to examine women's life trajectories at least 4 years after cancer diagnosis, and maximum 10 years after their diagnosis, which is the length of the follow-up in hospital services where recruitment will take place.

Exclusion Criteria:

* Does not speak French
* Under 18 years old
* Have been diagnosed with breast cancer before 2014 and after 2020

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women born in sub-Saharan Africa and in France who have been diagnosed with breast cancer between the 1st of January 2014 and the 31st of December 2020 and visiting three hospital (Saint-Louis University Hospital AP-HP; Delafontaine Hospital Saint-Denis; Robert Ballanger, Hospital, Aulnay-sous-Bois) in the greater Paris area.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Circumstances of breast cancer diagnosis | From first signs until breast cancer diagnosis, up to 10 years
  Proportion of women who declare, retrospectively, diagnosed following clinical signs, screening campaigns or medical prescription
Time between date of arrival in France and breast cancer diagnosis | From arrival in France until the date of diagnosis, up to 10 years
  Time to breast cancer diagnosis, from arrival in France, for women born in Sub-Saharan Africa
Time between breast cancer diagnosis and access to care | From date of diagnosis until date of first consultation for cancer care, and then each year up to 10 years
  Time between diagnostic and entry into breast cancer care (surgery, radiotherapy, chemotherapy, hormone therapy)
Breast cancer treatments | At time of diagnosis, and then each year up to 10 years
  Percentage of women who received surgery, radiotherapy, chemotherapy and/or hormone therapy as breast cancer treatment since diagnosis
Impact of the migration trajectory on access to breast cancer care | From arrival in France until breast cancer diagnosis, and then each year up to 10 after breast cancer diagnosis
  Percentage of undocumented women, women without health coverage after arrival in France and at the time of breast cancer diagnosis

SECONDARY OUTCOMES:
Breast cancer impact on sexuality | At time of diagnosis, and then each year up 10 years
  Proportion of women who declare, retrospectively, change in the frequency of sexual intercourse, sexual libido and in the intention to have a child since diagnosis
Impact of breast cancer and migration status on gender relations | At time of diagnosis, and then each year up to 10 years
  Proportion of women who declare, retrospectively, ongoing unions at the time of diagnosis, change in the ongoing union (strengthening, deterioration of unions), and proportion of women who declare, retrospectively, being supported by their partners following breast cancer diagnosis
Breast cancer impact on women's lives | At time of diagnosis, and then each year up to 10 years
  Proportion of women who report physical limitations following breast cancer diagnosis and treatments, and proportion of women who report being supported by someone other than their partner (for those who declare a partner) following breast cancer diagnosis
Impact of the disease on the professional situation | At time of diagnosis, and then each year up to 10 years
  Percentage of women employed at the time of diagnosis and then each year up to 10 years or at the time of data collection

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Robert Ballanger Hospital Aulnay-Sous-Bois, Aulnay-sous-Bois
  - Saint-Louis University Hospital AP-HP, Paris
  - Delafontaine Hospital Saint-Denis, Saint-Denis

REFERENCES:
- [Background] Anne Gosselin, Karna Coulibaly, Joseph Larmarange, Clémence Schantz. Plan de gestion des données du projet SENOVIE France. Institut de Recherche pour le Développement (IRD). 2024. ⟨hal-04563793⟩
- [Background] Louise Ludet, Luis Teixeira, Gaëtan des Guetz, Clémence Schantz, for the SENOVIE group. Therapeutic mobility and breast cancer in France: Experiences of African women. SSM - Qualitative Research in Health, Volume 4, 2023. https://doi.org/10.1016/j.ssmqr.2023.100314.
- [Derived] Coulibaly K, Schantz C, Teixeira L, Degrees du Lou A, Des Guetz G, Hocini H, Zelek L, Larmarange J, Gosselin A; SENOVIE study group; SENOVIE study group. A Life course approach to investigate breast cancer and migration in the greater Paris area: the SENOVIE study protocol. BMJ Open. 2025 Apr 2;15(4):e095759. doi: 10.1136/bmjopen-2024-095759. PMID 40180375
- See also: Data management plan — https://dmp.opidor.fr/plans/27712/export.pdf?export%5Bquestion_headings%5D=true